CLINICAL TRIAL: NCT05187637
Title: Analysis of the Application of a Patient Blood Management Program in Liver Transplantation Through Intravenous Iron Treatment in Patients on the Liver Transplant Waiting List
Brief Title: .Patient Blood Management Program in Liver Transplantation
Acronym: PBM-THO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Principal Investigator, Lourdes Pérez, Medical Doctor, Hospital Universitari de Bellvitge
Other Study IDs: EOM025/21
Record Dates: First submitted 2021-12-15; First posted 2022-01-12 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Iron Deficiency Anemia
Keywords: iron deficiency; liver transplantation; intravenous iron
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies | interventions — ferric carboxymaltose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention: Patients on the waiting list for liver transplantation with haemoglobin less than 11.5g/dL and transferrin saturation index less than 40% with ferritin less than 800mcg/L, which are considered iron deficiency susceptible to respond to intravenous iron administration.
  Interventions: Drug: intravenous iron
- Control: Patients on the waiting list for liver transplantation in the same period of the intervention cohort, with haemoglobin less than 11.5g/dL and transferrin saturation index more than 40%, which are considered of non susceptibles for iron supplement alone.

INTERVENTIONS:
Drug: intravenous iron — One dose of intravenous iron carboxymaltose calculated according to ganzoni's formula. If after thirty days of the first dose, a second dose of 500mg will be administered if the patient continues to meet the inclusion criteria.
  Other Names: ferinject
  Groups: Intervention

SUMMARY:
Transfusion management improvement programs, generally known as patient blood management (PBM) programs, are based on a set of perioperative measures aimed at improving clinical outcomes by avoiding unnecessary exposure to blood components.

In a recent series of liver transplants (LT) performed in Spanish centers belonging to the Spanish Liver Transplant Society, despite optimal hemostasis management and preservation of the vena cava, around 20% of patients required massive transfusion (considered as the administration of 6 or more red blood cell concentrates intraoperatively). In addition, 63% of the patients were transfused with at least one packed red cells during the operation.

By correcting the iron deficiency in patients who meet the criteria of the anemia study (transferrin saturation less than 20%), we could improve the hemoglobin level, which would allow a wider margin for the transfusion of red cell concentrates.

DETAILED DESCRIPTION:
This is a prospective observational multicenter study to evaluate the efficacy of iron administration in patients candidates to LT. Inclusion criteria Patients with Hb < 11.5 g/dL + and transferrin saturation index < 40%+ferritina <800mcg/L will receive Fe carboxymaltose iv* *Ganzoni formula modified (total iron dose = [actual body weight × (11.5-actual Hb)] × 2.4 + 500), and represent the intervention group. Those patients with Hb < 11.5 g/dL and transferrin saturation index > 40% will constitute the control group. The Intraoperative managed protocol was standardized within groups and Teams. Demographic and liver function test after iron administration will be registered; perioperative transfusion data will be recorded. Recruitment, treatment and follow-up will be conducted by monitored by an independent audit to assure the quality of data. Specific Data Unit not related to the participated Teams will do statistical analysis. The primary outcome is the feasibility of apply the first pillar of the patient blood management programs (PBM) in LT candidates. Secondary outcomes are the response rate (increase in Hb > 1 g/dL) to the intervention, and red blood cell requirements in both, intervention and control group

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis on the liver transplant waiting list
* haemoglobin lower than 11.5g/dL
* transferrin saturation index below 40%
* ferritin below 800mcg/L

Exclusion Criteria:

* refusal to participate
* Known hypersensitivity to Ferinject
* current infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis of the liver on the waiting list for liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-04-24 (Estimated); Study Completion 2023-04-24 (Estimated)

PRIMARY OUTCOMES:
degree of implementation of the PBM programme | 30 days after the intervention or pre-surgery
  To assess the degree of implementation of the PBM Programme in its first pillar in patients with iron deficiency anaemia, determining the degree and quality of implementation of the PBM programme in liver transplantation, measured as the percentage of patients complying with the iron correction protocol

SECONDARY OUTCOMES:
Effectiveness | Pre-surgery
  Percentage of responding patients, understanding positive response as an increase in haemoglobin ≥ 1 g/dl from inclusion in the study to the day of transplantation.
Clinical efficacy | immediately after the surgery
  Percentage of patients requiring transfusion and intraoperative massive transfusion and the number of red blood cell concentrates received per patient, compared to a cohort, adjusted for the characteristics of the included population, of patients transplanted in the same period with anaemia of inflammatory cause

OTHER OUTCOMES:
security | immediately after the intervention
  Safety variables related to iron administration.

CONTACTS AND LOCATIONS:
Overall Officials: Annabel MJ Blasi, MD, PhD, Study Director — Hospital Clinic Universitary
Locations (1):
- HUBellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided